CLINICAL TRIAL: NCT06102460
Title: The Effect of Pre-sleep Milk-derived Protein to Support Sleep Quality and Recovery in Elite Female Athletes
Brief Title: Pre-sleep Macros on Sleep Quality and Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: Milk Specialties Global (Industry)
Responsible Party: Principal Investigator, Michael J. Ormsbee, Director, Florida State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: STUDY00004409
Record Dates: First submitted 2023-10-13; First posted 2023-10-26 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Sleep
MeSH Terms: interventions — Carbohydrates

STUDY DESIGN:
Intervention Model Description: All participants will complete all 4 interventions with at least a 1 week wash out period in between.
Who Masked: Participant, Investigator
Masking Description: Neither the participant or investigator will know what treatment has been given until un-blinding at the completion of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Casein Protein (Active Comparator): Each participant will consume a serving of casein protein mix.
  Interventions: Dietary Supplement: Casein protein
- a-lactalbumin (Active Comparator): Each participant will consume a serving of a-lactalbumin protein mix.
  Interventions: Dietary Supplement: a-lactalbumin protein
- Carbohydrate (Active Comparator): Each participant will consume a serving of carbohydrate mix.
  Interventions: Dietary Supplement: Carbohydrate
- Placebo (Placebo Comparator): Each participant will consume a serving of a placebo mix.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Casein protein — 40 grams of casein protein powder mixed with 8-10 fl. oz. of water.
  Arms: Casein Protein
Dietary Supplement: a-lactalbumin protein — 40 grams of a-lactalbumin protein powder mixed with 8-10 fl. oz. of water.
  Arms: a-lactalbumin
Dietary Supplement: Carbohydrate — 40 grams of a carbohydrate powder mixed with 8-10 fl. oz. of water.
  Arms: Carbohydrate
Dietary Supplement: Placebo — Zero calorie, placebo powder mixed with 8-10 fl. oz. of water.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to assess the effect of eating before bed (2 hours after dinner, 30mins before bed) and the effects this has on sleep and recovery measures in elite female athletes.

Participants will be randomized to 4 possible groups in a double-blind randomized cross over design. Each group will ingest 40 grams of one of the following nutrients as a liquid shake for 3 consecutive nights:

1. Casein Protein
2. a-lactalbumin Protein
3. Carbohydrate
4. Placebo

There will be at least 1 week washout period between each intervention.

Sleep and recovery outcome measures will be obtained through a WHOOP 4.0 wearable healthy tracking device. Subjective sleep and recovery will be obtained through subjective questionnaires. Food will be logged by participants on intervention days. Blood glucose will be measured using continuous glucose monitors.

ELIGIBILITY:
Inclusion Criteria:

* NCAA Division I female athlete
* Wearing WHOOP 4.0 device for >3 months

Exclusion Criteria:

* Musculoskeletal injuries limiting participation in regular team practice.
* Cardiometabolic diseases limiting participation in regular team practice.
* Pre-diagnosed sleep condition that would negatively affect sleep quality or quantity (sleep apnea, restless leg syndrome, night-feeding syndrome)
* Allergy to any dietary supplement used in protocol - e.g., lactose intolerant.
* Use of sleep aids such as but not limited to, melatonin.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-01-23 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Sleep | Data obtained from device 12 hours after ingestion of supplement
  Sleep score determined by WHOOP 4.0 wearable device
Recovery | Data obtained from device 12 hours after ingestion of supplement
  Recovery score determined by WHOOP 4.0 wearable device

SECONDARY OUTCOMES:
Subjective sleep score | Data obtained 1-2 hours after after subject awakes
  Subjective sleep score obtained from questionnaire
Subjective recovery score | Data obtained 1-2 hours after after subject awakes
  Subjective sleep score obtained from questionnaire
Blood glucose control | Continuous (24hours/day) during intervention days/nights
  Using the continuous glucose monitor, participants blood glucose response throughout the day and night relative to regular meals and intervention will be observed.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Sports Sciences and Medicine - Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No